CLINICAL TRIAL: NCT04550221
Title: Randomized Controlled Trial of the Shauriana Intervention to Integrate PrEP, Sexual Health, and Mental Health Support for Gay, Bisexual, and Other Men Who Have Sex With Men in Kenya
Brief Title: The Shauriana Intervention for GBMSM in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susan Graham, Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00009441; R34MH118950 (NIH)
Record Dates: First submitted 2020-08-30; First posted 2020-09-16 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention
Keywords: preexposure prophylaxis; sexual health; mental health; behavioral intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Pilot study with 10 intervention participants followed by randomized controlled trial with 60 participants assigned to the intervention or to standard care.
Who Masked: Outcomes Assessor
Masking Description: Laboratory testing for PrEP drug levels will be conducted in a blinded fashion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Shauriana intervention is aimed at promoting sexual health and preventing HIV through a comprehensive prevention toolbox including PrEP. Components of this intervention are: four weekly in-person sessions with a trained peer intervention specialist; optional additional in-person or by phone check-ins after the in-person sessions are delivered; and optional monthly group sessions.
  Interventions: Behavioral: Shauriana
- Standard care (Active Comparator): Standard care includes clinic-based HIV counseling and testing, screening for symptoms of sexually transmitted infections (STI), and individual counseling about HIV prevention methods. Standard of care counseling for HIV prevention in Kenya includes general information about HIV transmission and discussions of risk reduction including condom use. PrEP counseling sessions focus on PrEP knowledge, adherence tips, and strategies to address adherence barriers.
  Interventions: Behavioral: Shauriana

INTERVENTIONS:
Behavioral: Shauriana — The components of this intervention are: four weekly in-person sessions with a trained peer intervention specialist; optional additional in-person or by phone check-ins after the in-person sessions are delivered; and optional monthly group sessions. The four in-person health education and coaching sessions will be delivered once per week, by trained peer facilitators who identify as GBMSM. These sessions will focus on the following topics: sexual health basics (understanding how HIV and STIs are transmitted, prevented, and diagnosed/treated), relationships (types of relationships we have, characteristics of healthy relationships, communication skills), stress and coping (understanding mental health challenges, adaptive and maladaptive coping strategies), and healthy sexuality and empowerment (understanding sexual orientation and gender identity, challenging stereotypes about GBMSM, making sexual choices).

SUMMARY:
The Shauriana intervention, developed from qualitative work using a community-based participatory approach, aims to integrate PrEP, sexual health, and mental health support for gay, bisexual, and other men who have sex with men in Kenya. This study consists of a brief pilot test phase with 10 participants, followed by a randomized, controlled trial with 60 participants.

DETAILED DESCRIPTION:
Gay, bisexual, and other men who have sex with men (GBMSM) are at high risk for HIV-1 acquisition, especially in rights-constrained settings such as Kenya, where men's access to HIV prevention has been impeded by homophobia, stigma, and discrimination. Pre-exposure prophylaxis (PrEP) has the potential to greatly reduce HIV acquisition risk in this key population if accessible, sustainable PrEP programming with tailored, effective adherence support can be provided. To this end, close collaboration between PrEP program implementers and GBMSM-led community-based organizations is essential. Based on preliminary qualitative work, this theory-based and culturally relevant PrEP support intervention is called Shauriana (Kiswahili for "we counsel each other"). The Shauriana intervention merges peer navigation and "integrated Next Step Counseling" (iNSC) to promote sexual health protection strategies, including PrEP uptake and adherence, among GBMSM in Kisumu. The present proposal aims to pilot the intervention among 10 participants for 3 months, and then to evaluate the Shauriana intervention for acceptability, feasibility, safety, and estimated effect on PrEP uptake and adherence, compared to standard of care, in a small randomized, controlled study with 60 participants followed for 6 months after enrollment. Results of the proposed research will have high impact by ensuring GBMSM involvement in the scale-up of effective PrEP programming for this key population in Kenya and providing a peer-led PrEP support model for GBMSM and other vulnerable and marginalized populations in African settings.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male at birth and identifies as male, according to self-report
* 18 to 35 years of age
* Resident in the Kisumu area for ≥12 months
* Reports anal intercourse with a man in the past 3 months
* Not currently taking PrEP for HIV prevention in the past 3 months
* Willing to provide complete locator information
* Willing to undergo all study procedures, including HIV testing and counselling
* Not currently participating in any HIV prevention or vaccine study
* Planning to remain in the study area for at least 6 months

For the pilot study only, men will be required to speak English, in order to expedite the study team's analysis of feedback from these participants in preparation for the randomized controlled trial (RCT). Of note, approximately 50%-60% of young MSM in Kisumu speak English.

Exclusion Criteria:

* Unable to understand the study purpose and procedures
* Unwilling to adhere to study procedures
* Currently under the influence of alcohol or drugs
* Prior diagnosis of HIV infection

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biologically male at birth and identifies as male, according to self-report
Enrollment: 63 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Graham, MD, MPH, PhD, Principal Investigator — University of Washington
Locations (1):
- Anza Mapema Clinic, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Study data will be available upon request after publication of the main study manuscripts. Researchers requesting access to data/resources will be asked to submit a request in writing describing their qualifications including their certification by their local IRB, analytic plans and other uses of the data/resources, and plans to secure the confidentiality and safety of the data. They will be required to agree in writing that they will not share the data with others, will use it only for the research purpose(s) delineated, and will return or destroy the data upon completion. In order to maintain protection of our participants' privacy, no directly identifying information will be shared with outside investigators. Given the sensitive nature of the data we are collecting, including HIV diagnosis and sexual risk behavior, we will not create a public access file.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After reporting of the trial results
Access Criteria: Data sharing agreement with study investigators

REFERENCES:
- [Result] Harper GW, Lewis KA, Norwitz GA, Odhiambo EO, Jadwin-Cakmak L, Okutah F, Lauber K, Aloo T, Collins B, Gumbe E, Amico KR, Olango K, Odero W, Graham SM. "God Didn't Make a Mistake in Creating Me": Intrapersonal Resilience Processes among Gay and Bisexual Male Youth in Kenya. Adolescents. 2021 Sep;1(3):267-282. doi: 10.3390/adolescents1030020. Epub 2021 Jul 13. PMID 35665057
- [Result] Jadwin-Cakmak L, Lauber K, Odhiambo EO, Collins B, Gumbe E, Norwitz GA, Aloo T, Lewis KA, Okutah F, Amico KR, Olango K, Odero W, Graham SM, Harper GW. "When you talk it out ... you will feel like the burden has somehow gone down, you will feel light": Social Support Received by Gay, Bisexual, and Other Men Who Have Sex with Men in Western Kenya. Int J Environ Res Public Health. 2022 Feb 1;19(3):1667. doi: 10.3390/ijerph19031667. PMID 35162690
- [Result] Graham SM, Okall DO, Mehta SD, Obondi E, Ng'ety G, Ochieng E, Jadwin-Cakmak L, Amico KR, Harper GW, Bailey RC, Otieno FO. Challenges with PrEP Uptake and Adherence Among Gay, Bisexual, and Other Men Who Have Sex with Men in Kisumu, Kenya. AIDS Behav. 2023 Apr;27(4):1234-1247. doi: 10.1007/s10461-022-03860-w. Epub 2022 Oct 11. PMID 36219270
- [Derived] Graham SM, Wang L, Jadwin-Cakmak L, Odhiambo EO, Bauman K, Okall D, Odero W, Otieno F, Amico KR, Harper GW. Acceptability, Feasibility, and Safety of the Shauriana Intervention for Young Kenyan Gay, Bisexual, and Other Men who Have Sex with Men, and Exploration of Potential Impact on Sexual Health Outcomes. AIDS Behav. 2025 Nov 25. doi: 10.1007/s10461-025-04965-8. Online ahead of print. PMID 41288881
- [Derived] Jadwin-Cakmak L, Harper GW, Ochieng E, Amico KR, Aloo T, Okutah F, Gumbe E, Olango K, Okall DO, Otieno FO, Odero W, Graham SM. Participatory development of the Shauriana program to integrate sexual health and mental health support for young gay and bisexual men and other men who have sex with men in Kenya. Adv Glob Health. 2025;4(1):2442813. doi: 10.1525/agh.2025.2442813. Epub 2025 Mar 6. PMID 40296878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening and enrollment took lace between May 10 and September 8 2021 at the Anza Mapema Clinic in Kisumu, Kenya. Overall, 71 individuals were screened, of whom 11 were not eligible. Sixty-three individuals were enrolled and completed a baseline visit.
Pre-assignment Details: Three individuals who were assigned to the intervention arm were withdrawn from the study after the baseline visit because they moved immediately from the study area or otherwise turned out not to be available for study and/or intervention visits.
Period: Overall Study
Arm/Group | Intervention | Standard Care
Started | 32 | 31
Month 1 Visit | 29 | 31
Month 3 Visit | 29 | 30
Month 6 Visit | 27 | 27
Exit Interviews | 28 | 0 (Exit interviews were only conducted for intervention participants.)
Completed | 27 | 27
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawn | 3 | 0
Not completed — Moved from the study area after receiving the intervention | 2 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis excludes the 3 intervention participants who were withdrawn immediately after the baseline visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard Care | Total
Number analyzed (Participants) | 29 | 31 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [22 to 27] | 26 [23 to 28] | 25 [22 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 31 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Kenyan | 29 | 31 | 60
Region of Enrollment [Number; unit: participants]
  Kenya | 29 | 31 | 60
Ever married to a female [Count of Participants; unit: Participants]
  No | 28 | 28 | 56
  Yes | 1 | 3 | 4
Education [Count of Participants; unit: Participants] — Highest level of education attained
  Participants
    Completed primary school | 1 | 2 | 3
    Completed secondary school | 18 | 15 | 33
    Completed certificate, diploma, or degree | 8 | 10 | 18
    Current student | 2 | 4 | 6
Sex of partners in past 3 months [Count of Participants; unit: Participants]
  Male only | 15 | 19 | 34
  Male and female | 14 | 12 | 26
Condom use last sex [Count of Participants; unit: Participants]
  Yes | 27 | 22 | 49
  No | 2 | 9 | 11

OUTCOME MEASURES:

1. Primary Outcome: Completion of Exit Interview
Description: All intervention arm participants were invited to provide qualitative feedback on intervention acceptability in an exit interview
Time Frame: Month 6
Population: Exit interviews only offered to intervention participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 28 | 0
Participants | 28 |

2. Primary Outcome: Intervention Feasibility
Description: Intervention session attendance
Time Frame: Month 6
Population: Intervention feasibility was only assessed in the intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 29 | 0
Participants
  Completed all 5 intervention sessions only | 11 | 0
  Completed all 5 intervention sessions plus an optional session | 18 | 0

3. Primary Outcome: Intervention Safety
Description: Adverse events reported by participants
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 29 | 31
Participants
  Adverse events reported | 0 | 0
  Adverse events not reported | 29 | 31

4. Secondary Outcome: PrEP Uptake
Description: Ongoing PrEP use (yes or no) assessed by ACASI
Time Frame: Month 1, Month 3, and Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 29 | 31
Participants
  Month 1: Used PrEP since last visit | 16 | 14
  Month 1: Did not use PrEP since last visit | 12 | 15
  Month 1: Missed visit or missing data | 1 | 2
  Month 3: Used PrEP since last visit | 17 | 18
  Month 3: Did not use PrEP since last visit | 11 | 12
  Month 3: Missed visit or missing data | 1 | 1
  Month 6: Used PrEP since last visit | 11 | 13
  Month 6: Did not use PrEP since last visit | 16 | 14
  Month 6: Missed visit or missing data | 2 | 4

5. Secondary Outcome: PrEP Adherence
Description: In the last 30 days, how good a job did you do at taking your PrEP daily?
Time Frame: Month 1, Month 3, and Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 29 | 31
Participants
  Month 1: Poor | 0 | 0
  Month 1: Fair | 0 | 1
  Month 1: Good | 5 | 7
  Month 1: Very good | 4 | 2
  Month 1: Excellent | 2 | 0
  Month 1: Missing or not taking PrEP | 18 | 21
  Month 3: Poor | 1 | 0
  Month 3: Fair | 2 | 7
  Month 3: Good | 5 | 6
  Month 3: Very good | 2 | 2
  Month 3: Excellent | 2 | 2
  Month 3: Missing or not taking PrEP | 17 | 14
  Month 6: Poor | 0 | 0
  Month 6: Fair | 1 | 3
  Month 6: Good | 4 | 3
  Month 6: Very good | 0 | 3
  Month 6: Excellent | 2 | 2
  Month 6: Missing or not taking PrEP | 22 | 20

6. Secondary Outcome: PrEP Drug Levels
Description: Tenofovir levels measured in dried blood spots
Time Frame: Month 3 and Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard Care
Number analyzed (Participants) | 29 | 31
Participants
  Month 3: TFV-DP detected | 3 | 7
  Month 3: TFV-DP not detected | 23 | 23
  Month 3: Missing | 3 | 1
  Month 6: TFV-DP detected | 4 | 6
  Month 6: TFV-DP not detected | 22 | 21
  Month 6: Missing | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 months, and focused on potential social harms of this sociobehavioral intervention.
Arm/Group | Intervention | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT04550221/Prot_SAP_ICF_000.pdf